CLINICAL TRIAL: NCT00003055
Title: Phase II Trial of Cisplatin and Irinotecan in Patients With Advanced Esophageal Cancer
Brief Title: Cisplatin and Irinotecan in Treating Patients With Locally Advanced or Metastatic Esophageal or Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-060; CDR0000065703 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1306
Record Dates: First submitted 1999-11-01; First posted 2004-07-30 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Irinotecan

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with locally advanced or metastatic esophageal or gastric cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate of combined cisplatin and irinotecan in patients with metastatic or locally advanced (inoperable or recurrent) esophageal or gastric cancer. II. Evaluate the toxic effects both qualitatively and quantitatively of cisplatin and irinotecan in these patients. III. Estimate the disease free and overall survival of these patients. IV. Assess whether the response proportion differs between squamous cell and adenocarcinoma of the esophagus. V. Evaluate quality of life issues using the Memorial Symptom Assessment Scale, the FACT-G questionnaire, and the dysphagia scale.

OUTLINE: Patients receive cisplatin and irinotecan on days 1, 8, 15, and 22 for 4 weeks, followed by a 2 week rest period. Each treatment course lasts 6 weeks. Patients receive at least 3 courses of therapy if the treatment is well tolerated and no disease progression is documented. Patients attaining a complete response receive additional courses of therapy at the discretion of the investigator. Tumor status is reassessed at 6 weeks and every 12 weeks thereafter. Patients are followed until death.

PROJECTED ACCRUAL: A total of 28-50 patients will be accrued within 12-18 months. Accrual for adenocarcinoma of the esophagus is complete.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locally advanced (surgically unresectable) or metastatic squamous cell of the esophagus or carcinoma of the stomach Patients with tumor extension below the GE junction into the proximal stomach must have the bulk of the tumor involve the esophagus or GE junction Bidimensionally measurable or evaluable disease No CNS metastases or carcinomatous meningitis No bone metastases (Closed to adenocarcinoma of the esophagus as of 05/1998)

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: Karnofsky 60-100% Life Expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 3 times upper limit of normal (ULN)(no greater than 5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No unstable angina No New York Heart Association class III or IV cardiac disease Pulmonary: No interstitial pulmonary fibrosis Other: Not pregnant or nursing Negative pregnancy test No active or uncontrolled infection No prior malignancy for at least 5 years, except: Nonmelanoma skin cancer Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior radiation to the pelvis Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-06; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States